CLINICAL TRIAL: NCT06270485
Title: Influence of Positive-End-Expiratory-Pressure (PEEP) on Cardiac Output in Mechanically Ventilated Children
Acronym: IPCOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jan Clausen, Dr. med. / MD, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA2/224/23
Record Dates: First submitted 2024-02-02; First posted 2024-02-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Ventilation Therapy; Complications; Congenital Heart Disease; Children, Only; Hemodynamic Instability
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ventilated children (Other): Application of different PEEP-levels during invasive mechanical ventilation
  Interventions: Procedure: PEEP

INTERVENTIONS:
Procedure: PEEP — Application of different PEEP-Levels during invasive mechanical ventilation

SUMMARY:
Interventional Trial to determine the Effect of different PEEP levels on Cardiac output and right-ventricular function in mechanically ventilated children < 5 years of age with congenital heart disease.

DETAILED DESCRIPTION:
Different PEEP-levels will be applied during invasive mechanical ventilation to describe Cardio-pulmonary interactions in children with congenital heart disease (CHD). An additional trial with the same study protocol is planned in a cohort of children with primarily pulmonary disease without CHD after completion of this trial. Esophageal pressure-monitoring, Ultrasound, respiratory mechanics and electrical impedance tomography will be used

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanical ventilation
* congenital heart disease (biventricular anatomy)

Exclusion Criteria:

* univentricular hearts
* ECMO/VAD

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | 1 year
  change in CO during intervention

SECONDARY OUTCOMES:
TAPSE (cm) | 1 year
  Excursion of the TV annulus
respiratory mechanics | 1 year
  Tidal Volume (ml/kg)
TAPSV (cm/s) | 1year
  systolic excursion of the TV annulus with tissue doppler
Global Strain RV (%/sec) | 1year
  shortening of the RV myocardium during systole
Lung Compliance (ml/Min/kg) | 1year
  compliance of lung tissue
Esophageal Pressure (mbar) | 1year
  monitoring with balloon
EIT | 1year
  Tidal Volume distribution

CONTACTS AND LOCATIONS:
Overall Officials: Jan Clausen, MD, Principal Investigator — Charité
Locations (2):
- Deutsches Herzzentrum der Charité, Berlin, State of Berlin, Germany
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] "Electrical impedance tomography during open heart surgery and on the cardiac icu is feasible to monitor ventilation in children with congenital heart disease" J.-C. Clausen, M. Emeis, M. Kleine-Brueggeney, M.-Y. Cho, M. Kneyber and O. Miera Intensive Care Medicine - Paediatric and Neonatal 2024 Vol. 2 Issue 1 Pages 19 DOI: 10.1007/s44253-024-00043-4
- [Derived] Clausen JC, Emeis M, Hollander R, Miera O, Kleine-Brueggeney M, Blokpoel RGT, Garfias-Veitl T, Asendorf T, Vadiunec VV, Photiadis J, Berger F, Kneyber MCJ. Effect of Positive End-Expiratory Pressure on Cardiac Index and Right Ventricular Performance in Ventilated Children Post-Cardiac Surgery. Pediatr Crit Care Med. 2026 Feb 1;27(2):176-186. doi: 10.1097/PCC.0000000000003880. Epub 2025 Dec 19. PMID 41416857